CLINICAL TRIAL: NCT05021640
Title: A Phase 1, Double-blind, Placebo-controlled, Single-ascending Dose, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Study of DCR-AUD in Healthy Volunteers
Brief Title: Study of DCR-AUD in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dicerna Pharmaceuticals, Inc., a Novo Nordisk company (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: DCR-AUD-101; U44AA027404 (NIH)
Record Dates: First submitted 2021-08-18; First posted 2021-08-25 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Alcohol Use Disorder (AUD)
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants, Investigators, site staff, the CRO staff, and the Sponsor Medical Monitor will be blinded to the randomization. Other members of the Sponsor staff will be unblinded for the duration of the study. Complete details will be presented in the Study Blinding Plan.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1: DCRAUD 80 mg (Experimental): Participant received a single dose of DCR-AUD 80 mg, subcutaneous injection on Day 1.
  Interventions: Drug: DCR-AUD
- Cohort 2: DCRAUD 240 mg (Placebo Comparator): Participant received a single dose of DCR-AUD 240 mg, subcutaneous injection on Day 1.
  Interventions: Drug: DCR-AUD
- Cohort 3: DCR-AUD 480 mg (Experimental): Participant received a single dose of DCR-AUD 480 mg, subcutaneous injection on Day 1.
  Interventions: Drug: DCR-AUD
- Cohort 4: DCR-AUD 960 mg (Placebo Comparator): Participant received a single dose of DCR-AUD 960 mg, subcutaneous injection on Day 1.
  Interventions: Drug: DCR-AUD
- Pooled Placebo (Experimental): Participant received a single dose of DCR-AUD matching placebo, subcutaneous injection on Day 1.
  Interventions: Drug: Placebo for DCR-AUD

INTERVENTIONS:
Drug: DCR-AUD — DCR-A1203, the drug substance of DCR-AUD, is a synthetic double-stranded (hybridized duplex) RNA oligonucleotide conjugated to GalNAc ligands that enable specific hepatic access and uptake after subcutaneous administration. DCR-AUD is a sterile solution of DCR-A1203 at a concentration of 160 mg/mL in water for injection (WFI).
  Other Names: DCR-A1203
  Arms: Cohort 1: DCRAUD 80 mg; Cohort 2: DCRAUD 240 mg; Cohort 3: DCR-AUD 480 mg; Cohort 4: DCR-AUD 960 mg
Drug: Placebo for DCR-AUD — 0.9% saline for injection
  Other Names: Placebo
  Arms: Pooled Placebo

SUMMARY:
DCR-AUD will be evaluated for safety, tolerability, pharmacokinetics, and pharmacodynamics in healthy volunteers.

DETAILED DESCRIPTION:
DCR-AUD is being developed for the treatment of alcohol use disorder (AUD) in adults using an RNA interference (RNAi) technology platform. This is a 24-week, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, PK, and PD of single-ascending doses (SAD) of DCR-AUD administered to adult HVs. The single doses of DCR-AUD will be administered to adult HVs across 4 sequential cohorts (3 planned [80 mg, 240 mg, 480 mg] and one optional [960 mg]). Each cohort will comprise a sentinel group of 3 participants (2 active, 1 placebo) and an expanded group of 6 participants (4 active, 2 placebo). The sentinel group will be followed for the assessment of safety and tolerability and characterization of PK but who will not undergo any EIAs. Participants will receive a single dose of study intervention on Day 1 and will be followed for 24 weeks. Participants who have positive ethanol reaction symptoms at the Day 169 EIA (e.g., nausea, vomiting, or substantial flushing) will return every 28 (±7) days for follow-up EIAs until the positive ethanol reaction symptoms abate. These conditional follow-up (CFU) EIAs will not require overnight admission to the clinic, but all other aspects of the EIA will be conducted (see Table 3). Participants will be observed for not less than 6 hours after ethanol administration and will not be discharged until the Investigator deems it medically safe to do so.

ELIGIBILITY:
Inclusion criteria

* Male and female participants, between 21 and 65 years of age (inclusive), who were social drinkers of modest amounts of alcohol (less than or equal to (≤) 2 drinks/day, ≤ 3 days/week) and would be able to refrain from drinking alcohol during the outpatient portion of the trial
* Overtly healthy, as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* Negative screen for drugs of abuse (to include at minimum: amphetamines, barbiturates, cocaine, opioids, and benzodiazepines) at Screening and Day 1. Cannabis will not be recorded as a drug of abuse for this study.
* Had a negative test for Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV-2) infection on Day -1 and prior to admission to the clinical unit.
* Systolic BP in the range of 90 to 140 millimetre(s) of mercury (mmHg) and diastolic BP in the range of 50 to 95 mmHg, and body mass index (BMI) within the range of 18.0 to 32.0 kilogram per square meter (kg/m^2) (inclusive).

Exclusion Criteria:

* History of any medical condition that may interfere with the absorption, distribution, or elimination of study intervention, or with the clinical and laboratory assessments in this study, including (but not limited to): chronic or recurrent renal disease, functional bowel disorders (e.g., frequent diarrhea or constipation), clinically significant cardiovascular or pulmonary disease or has cardiovascular or pulmonary disease requiring pharmacologic medication, GI tract disease, pancreatitis, seizure disorder, mucocutaneous, or musculoskeletal disorder.
* Any history of severe or recent clinically significant depression, anxiety, bipolar disorder, schizophrenia, or other neuropsychiatric disorder that, in the judgment of the Investigator, represents a safety risk to the individual were they to participate in the trial
* History of delirium tremens or alcohol-related seizures.
* History of significant adverse reaction(s) to alcohol.
* History of substance use disorder (SUD), including alcohol (AUD) or illicit drug use (excluding cannabis) within the preceding 12 months. Nicotine use is permitted.
* History of any concomitant medical condition for which alcohol consumption is prohibited or advised against by the participant's physician or health care provider.
* History of multiple drug allergies or a history of allergic reaction to an oligonucleotide based therapy

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Parexel Los Angeles Early Phase Clinical Unit, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this trial 36 healthy participants were randomized to four ascending-dose cohorts (80 milligram [mg], 240 mg, 480 mg, 960 mg) and placebo.
Groups:
- Cohort 1: DCR-AUD 80 mg: Participant received a single dose of DCR-AUD 80 mg, subcutaneous injection on Day 1.
- Cohort 2: DCR-AUD 240 mg: Participant received a single dose of DCR-AUD 240 mg, subcutaneous injection on Day 1.
Period: Overall Study
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg | Pooled Placebo
Started | 6 | 6 | 6 | 6 | 12
Safety Population | 6 | 6 | 6 | 6 | 12
Pharmacodynamic Population | 4 | 4 | 4 | 4 | 8
Completed | 6 | 6 | 6 | 6 | 11
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants randomly assigned to study intervention and who received the full dose of study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg | Pooled Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 12 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (10.29) | 36.3 (12.26) | 34.2 (14.44) | 32.8 (4.88) | 41.3 (12.19) | 39.6 (12.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 4 | 8 | 24
  Male | 3 | 2 | 1 | 2 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 2 | 4 | 3 | 14
  Not Hispanic or Latino | 4 | 3 | 4 | 2 | 9 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 1 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 1 | 3 | 7
  White | 5 | 4 | 4 | 3 | 8 | 24
  More than one race | 0 | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An Adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. A TEAE is defined as an AE that begins or that worsens in severity after the study drug has been administered. An SAE is defined as any untoward medical occurrence that at any dose: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, leads to a congenital anomaly /birth defect, is the other important medical event.
Time Frame: From Day 1 up to 24 Weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg | Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
Participants
  TEAEs | 4 | 5 | 4 | 2 | 9
  SAEs | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Severity Grades of TEAEs
Description: An AE is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A TEAE is defined as an AE that begins or that worsens in severity after the study drug has been administered. As per the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0, Grade 1: mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; treatment not indicated; Grade 2: moderate; minimal, local, or noninvasive treatment indicated; limiting age-appropriate activities of daily living; Grade 3: severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care activities of daily living; Grade 4: life-threatening consequences; urgent treatment indicated; Grade 5: fatal.
Time Frame: From Day 1 up to 24 Weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg | Pooled Placebo
Number analyzed (Participants) | 4 | 5 | 4 | 2 | 9
Participants
  Grade 1 | 4 | 5 | 4 | 2 | 9
  Grade 2 | 2 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLTs) as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0
Description: DLT is defined as an AE of greater than or equal to (>=) Grade 3 intensity (CTCAE Version 5.0) in one participant, unless it is clearly the result of a non-study-related event OR any 2 AEs of >= Grade 2 intensity in the same body system in one participant.
Time Frame: From Day 1 up to 24 Weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg | Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
Participants | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Change From Baseline in Clinically Significant Abnormal Vital Signs
Description: Number of participants with change from baseline in clinically significant abnormal vital signs (temperature, pulse rate, respiratory rate, and blood pressure) is presented.
Time Frame: From Baseline (Day -1) up to 24 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg | Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
Participants | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Change From Baseline in Clinically Significant Abnormal Electrocardiogram (ECG) Findings
Description: Number of participants with change from baseline in clinically significant abnormal ECG findings (Heart rate, PR interval, QRS interval, QT interval and QT interval using Fridericia's correction [QTcF]) is presented.
Time Frame: From Baseline (Day -1) up to 24 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg | Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
Participants | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Change From Baseline in Clinically Significant Abnormal Laboratory Values
Description: Number of participants with change from baseline in clinically significant abnormal laboratory values (hematology, clinical chemistry, coagulation and routine urinalysis parameters) is presented.
Time Frame: From Baseline (Day -1) up to 24 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg | Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
Participants | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Change From Baseline in Clinically Significant Physical Examination Findings
Description: Number of participants with change from baseline in clinically significant physical examination findings (assessments of the cardiovascular, respiratory, gastrointestinal, neurological, and skin systems and inspection of the injection site) is presented.
Time Frame: From Baseline (Day -1) up to 24 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg | Pooled Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
Participants | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: AUC0-last: Area Under the Plasma Concentration Curve From Time Zero to the Last Quantifiable Concentration of DCR-AUD
Description: AUC0-last is defined as the area under the plasma concentration curve from time zero to the last quantifiable concentration of DCR-AUD.
Time Frame: Day 1: Predose, at 15 and 30 minutes, 1, 2, 4, 6, 8, 24, 48, 72 hours post dose; Day 15: Once Post dose
Population: Pharmacokinetic (PK) analysis population included all participants randomly assigned to study intervention and who received a full dose of DCR-AUD and had sufficient data for at least 1 postdose PK assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram per millilitre (h*ng/mL)
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour*nanogram per millilitre (h*ng/mL) | 5710 (25.2) | 19300 (18.8) | 49000 (26.9) | 106000 (29.3)

9. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration of DCR-AUD
Description: Cmax is defined as maximum observed plasma concentration of DCR-AUD during a dosing interval.
Time Frame: Day 1: Predose, at 15 and 30 minutes, 1, 2, 4, 6, 8, 24, 48, 72 hours post dose; Day 15: Once Post dose
Population: PK analysis population included all participants randomly assigned to study intervention and who received a full dose of DCR-AUD and had sufficient data for at least 1 postdose PK assessment.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per millilitre (ng/mL)
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
nanogram per millilitre (ng/mL) | 371 (20.4) | 956 (26.3) | 2580 (46.1) | 5350 (51.3)

10. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration of DCR-AUD (Cmax)
Description: Tmax is defined as time to reach the maximum plasma concentration (Cmax) of DCR-AUD.
Time Frame: Day 1: Predose, at 15 and 30 minutes, 1, 2, 4, 6, 8, 24, 48, 72 hours post dose; Day 15: Once Post dose
Population: as for outcome 9
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
hours | 4.00 [0.50 to 8.22] | 7.17 [1.15 to 8.02] | 4.05 [1.13 to 8.03] | 6.00 [0.65 to 8.12]

11. Secondary Outcome: t1/2: Apparent Terminal Elimination Half-life of DCR-AUD
Description: t1/2 is defined as apparent terminal elimination half-life of DCR-AUD.
Time Frame: Day 1: Predose, at 15 and 30 minutes, 1, 2, 4, 6, 8, 24, 48, 72 hours post dose; Day 15: Once Post dose
Population: PK analysis population included all participants randomly assigned to study intervention and who received a full dose of DCR-AUD and had sufficient data for at least 1 postdose PK assessment. Here, Overall Number of Participants Analyzed" signifies participants with available data for this outcome measure.
Measure: Median (Full Range); unit: hours
Groups:
- Cohort: DCR-AUD 80 mg: Participant received a single dose of DCR-AUD 80 mg, subcutaneous injection on Day 1.
Arm/Group | Cohort: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg
Number analyzed (Participants) | 3 | 4 | 2 | 1
hours | 7.67 [6.26 to 8.74] | 7.62 [6.35 to 8.84] | NA [4.67 to 5.82] — Median is not calculable due to two participants with data | NA [35.4 to 35.4] — Median is not calculable due to one participant with data

12. Secondary Outcome: Fe%0-72: Urinary Cumulative Excretion as % of Unchanged DCR-AUD up to 72 Hours
Description: Urinary cumulative excretion as % of DCR-AUD at each interval collection (0- 4 hours, 0- 8 hours, 0-12 hours, 0-24 hours, 0-48 hours, 0-72 hours) is reported in this outcome measure.
Time Frame: At time interval between 0- 4 hours, 0- 8 hours, 0-12 hours, 0-24 hours, 0-48 hours, 0-72 hours
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of unchanged DCR-AUD
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
percentage of unchanged DCR-AUD
  Fe%0-4 | 1.47 (38.1) | 2.51 (32.9) | 4.23 (24.7) | 3.85 (28.9)
  Fe%0-8 | 7.22 (38.2) | 8.68 (26.8) | 10.8 (42.4) | 10.4 (39.2)
  Fe%0-12 | 12.8 (26.8) | 12.8 (27.2) | 17.6 (28.5) | 19.2 (33.5)
  Fe%0-24 | 24.6 (17.0) | 23.6 (43.9) | 35.2 (21.9) | 35.6 (32.6)
  Fe%0-48 | 28.8 (18.1) | 28.5 (40.8) | 41.6 (13.7) | 43.7 (20.5)
  Fe%0-72 | 28.9 (18.1) | 28.9 (40.6) | 42.2 (12.6) | 45.1 (19.4)

13. Secondary Outcome: CLR: Renal Clearance of the DCR-AUD From Plasma
Description: Renal clearance of the DCR-AUD from plasma is reported in this outcome measure.
Time Frame: Day 1: 0-4, 4-8, 8-12, 12-24, 24-48, and 48-72-hours post-dose
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/h)
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg
Number analyzed (Participants) | 6 | 6 | 6 | 6
Liter per hour (L/h) | 3760 (13.5) | 3590 (27.1) | 4170 (27.8) | 4180 (25.0)

14. Secondary Outcome: Six Symptom Responses During Ethanol Interactions Assessments (EIAs)
Description: The degree of aldehyde dehydrogenase 2 (ALDH2) reduction was measured by quantitative assessment of 6 symptom (flushing, headache, palpitations, light-headedness, nausea, and vomiting) responses during EIAs. Each of 6 symptoms was assessed at each of the 4 time points during each EIA. Composite score at each time point was the sum of severity ratings for each of the 6 symptoms. Peak composite score (of the 3 post-alcohol initiation composite scores at each EIA test) was used as the subject's peak score for that EIA test. The point system was as follows: 0 point = symptom not present, 1 point = mild severity of symptom, 2 points = moderate severity of symptom and 3 points = severe severity of symptom. Participants were given a composite score, which was the sum of the scores of all 6 symptoms (highest possible score is 18).
Time Frame: Day -1, Day 4, Day 15, Day 29, Day 57, Day 85, Day 113 and Day 169
Population: Pharmacodynamic population (PP) included all participants randomly assigned to study intervention and who received a full dose of study intervention and had sufficient data for at least 1 postdose pharmacodynamic (PD) assessment. Here, number analysed signifies participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg | Pooled Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 8
score on a scale
  Day -1 | 0.8 (0.96) | 1.3 (1.50) | 1.0 (1.41) | 0.3 (0.50) | 0.3 (0.46)
  Day 4 | 1.0 (1.15) | 0 (0) | 0.8 (1.50) | 0.3 (0.50) | 0.4 (0.52)
  Day 15: number analyzed (Participants) | 4 | 4 | 3 | 4 | 7
  Day 15 | 0.5 (0.58) | 0.3 (0.50) | 0 (0) | 0 (0) | 0.3 (0.76)
  Day 29 | 0.8 (0.96) | 0 (0) | 0 (0) | 0.5 (1.00) | 0.3 (0.71)
  Day 57 | 0.3 (0.50) | 0 (0) | 0 (0) | 0 (0) | 0.1 (0.35)
  Day 85: number analyzed (Participants) | 3 | 4 | 4 | 4 | 6
  Day 85 | 0.3 (0.58) | 1.0 (1.41) | 0 (0) | 0 (0) | 0 (0)
  Day 113: number analyzed (Participants) | 4 | 4 | 4 | 4 | 6
  Day 113 | 0.5 (0.58) | 0.5 (1.00) | 0 (0) | 0 (0) | 0.2 (0.41)
  Day 169: number analyzed (Participants) | 4 | 4 | 4 | 4 | 7
  Day 169 | 0 (0) | 0.5 (1.00) | 0 (0) | 0 (0) | 0.3 (0.49)

15. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration of Acetaldehyde
Description: Maximum plasma concentration of acetaldehyde was measured to evaluate the pharmacodynamic effects of ALDH2 reduction by DCR-AUD during serial EIAs days.
Time Frame: Day -1, Day 4, Day 15, Day 29, Day 57, Day 85, Day 113 and Day 169
Population: Pharmacodynamic Population (PP) included all participants randomly assigned to study intervention and who received a full dose of study intervention and had sufficient data for at least 1 postdose PD assessment.
Measure: Mean (Standard Deviation); unit: micromolar (μM)
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg | Pooled Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 8
micromolar (μM)
  Day -1 | 33.7 (13.5) | 26.7 (15.3) | 11.3 (6.91) | 15.4 (8.45) | 29.4 (48.6)
  Day 4 | 30.9 (8.23) | 31.8 (24.2) | 10.3 (4.52) | 21.8 (13.8) | 31.9 (37.6)
  Day 15 | 8.11 (12.5) | 6.52 (4.57) | 11.9 (11.2) | 11.0 (5.31) | 20.4 (28.2)
  Day 29 | 13.4 (12.5) | 18.2 (8.31) | 25.6 (11.8) | 16.2 (9.48) | 10.6 (14.9)
  Day 57 | 16.4 (8.38) | 18.6 (6.56) | 31.0 (14.9) | 22.3 (6.34) | 18.6 (23.3)
  Day 85 | 12.8 (2.22) | 13.2 (4.87) | 26.5 (12.7) | 18.0 (4.30) | 8.38 (4.19)
  Day 113 | 20.6 (7.63) | 15.5 (4.91) | 23.3 (15.5) | 27.0 (12.6) | 14.8 (14.7)
  Day 169 | 11.8 (3.51) | 23.5 (12.2) | 31.9 (17.5) | 13.5 (7.09) | 15.8 (28.1)

16. Secondary Outcome: AUC0-2.5: Area Under the Concentration Time Curve From Time 0 to Fixed Time 2.5 of Acetaldehyde
Description: Area under the concentration time curve from time 0 to fixed time 2.5 of acetaldehyde was measured to evaluate the pharmacodynamic effects of ALDH2 reduction by DCR-AUD during serial EIAs days.
Time Frame: Day -1, Day 4, Day 15, Day 29, Day 57, Day 85, Day 113 and Day 169
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: hour*nanomolar (h*uM)
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg | Pooled Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 8
hour*nanomolar (h*uM)
  Day -1 | 44.4 (14.7) | 42.2 (27.2) | 10.3 (7.30) | 14.2 (11.5) | 39.1 (70.3)
  Day 4 | 41.8 (18.4) | 48.4 (31.9) | 8.29 (7.04) | 24.2 (22.4) | 41.6 (55.9)
  Day 15 | 4.18 (5.68) | 5.76 (3.95) | 11.7 (10.3) | 12.0 (9.88) | 21.3 (27.2)
  Day 29 | 10.4 (10.2) | 24.9 (15.7) | 33.0 (13.6) | 23.9 (12.7) | 13.7 (23.0)
  Day 57 | 25.3 (16.4) | 23.2 (11.2) | 32.6 (10.9) | 33.7 (13.1) | 25.9 (38.8)
  Day 85 | 18.5 (9.05) | 14.8 (8.94) | 36.5 (19.4) | 28.2 (6.83) | 9.06 (5.49)
  Day 113 | 28.0 (8.51) | 24.6 (13.4) | 28.6 (19.4) | 47.7 (23.3) | 21.7 (26.1)
  Day 169 | 13.1 (4.74) | 37.7 (25.4) | 42.2 (17.8) | 21.1 (7.51) | 21.0 (39.8)

17. Secondary Outcome: Change From Baseline in Heart Rate
Description: Heart rate is measured to evaluate the PD effects of ALDH2 reduction by DCR-AUD during serial EIA. Heart rate was monitored by telemetry during the EIAs.
Time Frame: Baseline (Day -1), Day 169
Population: Pharmacodynamic Population (PP) included all participants randomly assigned to study intervention and who received a full dose of study intervention and had sufficient data for at least 1 postdose PD assessment. Here, Overall Number of Participants Analyzed" signifies participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg | Pooled Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 7
beats/min | 10.0 (1.83) | 17.0 (10.23) | 13.0 (3.65) | 11.5 (11.47) | 18.4 (16.22)

18. Secondary Outcome: Change From Baseline in Facial Skin Temperature
Description: Change in facial skin temperature was measured to evaluate the PD effects of ALDH2 reduction by DCR-AUD during serial EIAs for the expanded group. Facial skin temperature was measured using a surface scanning thermometer.
Time Frame: Baseline (Day -1), Day 169
Population: Pharmacodynamic Population (PP) included all participants randomly assign ed to study intervention and who received a full dose of study intervention and had sufficient data for at least 1 postdose PD assessment. Here, Overall Number of Participants Analyzed" signifies participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: degree celsius
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg | Pooled Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 7
degree celsius | 0.55 (0.351) | 0.48 (0.330) | 0.28 (0.655) | 0.53 (0.250) | 0.51 (0.398)

19. Secondary Outcome: Change From Baseline in Subjective Effects of Alcohol Scale (SEAS) Score
Description: Subjective feelings of alcohol intoxication or intolerance is measured to evaluate the PD effects of ALDH2 reduction by DCR-AUD during serial EIAs. Participants' subjective experience of the effects of alcohol was assessed using the SEAS. The SEAS is a 14-item tool that allows participants to rate the subjective effects of alcohol. Participants rated the extent to which they were feeling (high/low arousal positive: relaxed, wobbly, lively, secure, woozy, fun, calm, dizzy, mellow, funny, talkative and high/low arousal negative: demanding, rude and aggressive) on an 11-point scale from (0 = not at all, 10 = extremely). higher values represent more effects.
Time Frame: Baseline (Day -1), Day 169
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort 4: DCR-AUD 960 mg | Pooled Placebo
Number analyzed (Participants) | 4 | 4 | 4 | 4 | 8
score on a scale
  High Arousal Negative | -0.335 (0.6700) | 1.333 (2.6650) | 0.915 (1.6175) | -0.083 (0.1650) | 0 (0.6157)
  High Arousal Positive | 0.938 (1.2311) | 1.250 (3.2404) | 0.313 (0.4732) | -1.125 (0.8539) | 0.438 (1.9491)
  Low Arousal Negative | 1.083 (2.5766) | 2.500 (1.5533) | 2.750 (3.1806) | 0.168 (1.4781) | -0.543 (1.4111)
  Low Arousal Positive | 0.688 (0.6575) | 0.500 (1.3540) | 0 (0) | 0.313 (0.5543) | 0.406 (0.5165)

ADVERSE EVENTS:
Time Frame: From Day 1 until end of the study (24 weeks).
Description: Safety population included all participants randomly assigned to study intervention and who received the full dose of study intervention. All serious and non-serious adverse events presented here are treatment emergent adverse events.
Groups:
- Cohort :4 DCR-AUD 960 mg: Participant received a single dose of DCR-AUD 960 mg, subcutaneous injection on Day 1.
Arm/Group | Cohort 1: DCR-AUD 80 mg | Cohort 2: DCR-AUD 240 mg | Cohort 3: DCR-AUD 480 mg | Cohort :4 DCR-AUD 960 mg | Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 4/6 | 5/6 | 4/6 | 2/6 | 9/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: DCR-AUD 80 mg (N=6) | Cohort 2: DCR-AUD 240 mg (N=6) | Cohort 3: DCR-AUD 480 mg (N=6) | Cohort :4 DCR-AUD 960 mg (N=6) | Pooled Placebo (N=12)
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0 | 2
Headache (Nervous system disorders) | 2 | 0 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 4 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 1 | 1 | 1 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1 | 0 | 2
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
SPONSOR agrees that the Principal Investigator shall have the right to publish or permit the publication of any information or material relating to or arising out of the work after prior submittal to SPONSOR provided that if SPONSOR shall so request, the investigator will delay publication for a maximum of ninety (90) days after submittal to SPONSOR to enable SPONSOR to protect its rights. SPONSOR will comment on such documents within thirty (30) days.

DOCUMENTS (2):
  • Study Protocol (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT05021640/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT05021640/SAP_001.pdf